CLINICAL TRIAL: NCT05943743
Title: Hiccups and Obstacles Of E-Learning Among Medical Students; A Cross-sectional Survey From Pakistan
Brief Title: Hiccups and Obstacles Of E-Learning Among Medical Sudents
Status: Recruiting | Type: Observational
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Rabia Khan, Assistant Professor, Bahria University
Other Study IDs: ERC 115/2022
Record Dates: First submitted 2023-03-16; First posted 2023-07-13 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Covid-19; E-learning; Medical Student
Keywords: Covid-19; obstacles; Screen Time
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Google form — * Self-administrated Questionnaire will be used for online survey. A pilot study was conducted on 30 sample size to check the reliability of questionnaire via statistical test.
  * A Five-point Likert scale (strongly disagree, disagree somewhat, Neutral, agree somewhat, strongly agree)

SUMMARY:
The COVID-19 Pandemic is the characterizing worldwide wellbeing emergency within recent memory. Since its development in Asia before the end of last year, the infection has spread to each mainland with the exception of Antarctica. Countries are dashing to moderate the spread of the illness by testing and treating patients, completing contact following, restricting travel, isolating residents, and dropping huge social occasions like games, shows, and educational institutes.

As almost every institution was closed for the safety of human kind. All educational institutes were also closed for any kind of education. Also, In Pakistan all educational institutes were closed since march 2020. It was impossible to keep educational activities closed for long. In order to keep educational activities in working e-learning was introduced through out the world. As many other countries Pakistan also started e-learning for all students.

DETAILED DESCRIPTION:
A world is transitioning from physical classes to hybrid studies. Pakistan is listed among third world country the availability of infra structure for hybrid study is not well developed, as consequence many hurdles and barriers are being faced by students, this has also been seen during covid-19 too. Distance E-learning in medical education may represent a suitable alternative to traditional learning to deliver high-quality education. The availability of essential infrastructures and efficient institutional strategies represent a major challenge for integrating distance learning in medical education.

During the pandemic, instructors and teaching staff were required to adapt quickly to the rapid transition in the education process and depend completely on the online platforms available, to deliver their courses, exams, and other required teaching and learning activities. While rapid transition to distance online learning was a mandatory and necessary action to ensure the learning continuity during the COVID-19 pandemic, it was not always a smooth process, that posed many challenges for instructors, learners.

Distance E-Learning is defined as using technology to deliver training, including technology supported learning either online, offline, or both. It is aimed at the effective construction of knowledge regarding individual experience, practice, and knowledge of the learners and students. Internet-based learning, computer-based learning, virtual classrooms, and digital collaboration all represent different types of e-learning

ELIGIBILITY:
Inclusion Criteria:

All undergraduate medical students of Pakistan.

Exclusion Criteria:

Postgraduate Medical students Teaching Faculty

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Undergraduate students of both private and government sector of medical institutes.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Difference of students educational level will assessed using Likert scale | 30 days
  During lockdown due to covid-19 medical students studies effected drastically. Academic level will be measured through likert scale in which 1 means good, 2 means average and 3 means below average. Academic level will be compared on the basis of students reply before and during covid academic result.

SECONDARY OUTCOMES:
Majority of students are facing internet and accessibility problems during online classes | 30 days
  students problem during online classes assessed using likert scale in which 1 means minimum issues facing and 5 means maximum issues facing during online classes

OTHER OUTCOMES:
Level of interest among students were very low due to online classes | 30 days
  Interest level towards studies was low may be due to technical issues. these parameters will be assessed through Likert Scale, in which 1 means strongly agree, 2 means agree, 3 means neutral, 4 mean disagree and 5 means strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Khan, Msc(PT), Principal Investigator — Bahria University
Locations (1):
- BUMDC, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data collection procedure, results and limitation and strengths will be shared through publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: By the end of year 2023
Access Criteria: Publications